CLINICAL TRIAL: NCT02586792
Title: Phase II, Open-Label Study of the Safety, Reactogenicity, and Immunogenicity of a Single Intramuscular Dose of Inactivated Influenza A/H7N9 Vaccine After Priming With Inactivated Influenza A/H7N7 Vaccine
Brief Title: H7N9 Boost in Healthy Adults
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 13-0044; Daughter study of 07-0023; HHSN272200800002C
Record Dates: First submitted 2015-10-22; First posted 2015-10-26 (Estimated); Last update posted 2018-08-22 (Actual); Status verified 2016-04

CONDITIONS: Influenza
Keywords: Influenza,Open-Label, Vaccine, Intramusclar, H7N7, H7N9, Non-adjuvanted, sub-study
MeSH Terms: conditions — Influenza, Human; Influenza in Birds

ARMS (2):
- Group 2 (Experimental): N up to 10 in prior receipt of a placebo in DMID Protocol 07-0023 will receive 45 mcg of HA/0.75 ml of Monovalent inactivated influenza A/H7N9 virus vaccine
  Interventions: Biological: Monovalent influenza A/H7N9 virus vaccine
- Group 1 (Experimental): N up to 40 in prior receipt of a monovalent inactivated influenza A/H7N7 virus vaccine in DMID Protocol 07-0023 will receive 45 mcg of HA/0.75 ml of Monovalent inactivated influenza A/H7N9 virus vaccine
  Interventions: Biological: Monovalent influenza A/H7N9 virus vaccine

INTERVENTIONS:
Biological: Monovalent influenza A/H7N9 virus vaccine — Monovalent influenza A/H7N9 virus vaccine.

SUMMARY:
The study will be an open-label phase 2 clinical trial of a single dose of an inactivated H7N9 influenza vaccine (non-adjuvanted). The subjects of the study will have previously participated in DMID trial 07-0023, evaluating inactivated Influenza A/H7N7 vaccine. In the previous study healthy adults 18 to 40 years old were randomized to receive two doses, 28 days apart, of placebo or 7.5, 15, 45, or 90 ug of the influenza vaccine by IM injection in a 1:1 ratio (N=25/vaccine group and 25 in placebo group). The primary objectives are to 1) assess the safety and reactogenicity of a single dose A/H7N9 vaccine in individuals who previously received two IM doses of an A/H7N7 vaccine or are A/H7 vaccine-naïve and 2) To assess the serum hemagglutination inhibition (HAI) antibody responses against A/H7N9 approximately 28 days following receipt of a single dose of A/H7N9 vaccine in individuals who previously received two IM doses of A/H7N7 vaccine or are A/H7 vaccine-naïve.

DETAILED DESCRIPTION:
This is a Phase II, open-label study in up to 50 males and non-pregnant females, 19 to 50 years old, inclusive, who are in good health and meet all entry criteria. The study is designed to assess the safety, reactogenicity, and immunogenicity of a single dose of a monovalent inactivated influenza A/H7N9 virus vaccine (45 mcg of HA/0.75 mL) manufactured by Sanofi Pasteur administered to healthy adults who previously received two doses of monovalent inactivated influenza A/H7N7 virus vaccine manufactured by Sanofi Pasteur or one or two doses of placebo in Protocol 07-0023. All subjects will receive a single dose of the inactivated influenza A/H7N9 vaccine delivered intramuscularly. Reactogenicity will be measured by the occurrence of solicited injection site and systemic reactions from the time of the study vaccination Day 1/Visit 01 through 8 days after the study vaccination. Unsolicited non-serious adverse events (AEs) will be collected from the time of the study vaccination through roughly 28 days after the study vaccination. Serious adverse events (SAEs) and new-onset chronic medical conditions will be collected from the time of the study vaccination through roughly 6 months after the study vaccination. Immunogenicity testing against A/H7N9 and A/H7N7 antigens will include performing hemagglutination inhibition (HAI) and neutralizing (Neut) antibody assays on serum obtained immediately prior to the study vaccination, and roughly 8 and 28 days after the study vaccination.

An additional 60 mL of venous blood will be drawn immediately prior to the study vaccination, and roughly 8 and 28 days after the study vaccination for exploratory cellular immunology assays.

The duration of this study for each subject will be roughly 6 months. The primary objectives are 1. to assess the safety and reactogenicity of a single dose monovalent inactivated influenza A/H7N9 virus vaccine in individuals who previously received two intramuscular doses of a monovalent inactivated influenza A/H7N7 virus vaccine or are A/H7 vaccine-naïve. 2. To assess the serum hemagglutination inhibition (HAI) antibody responses against A/H7N9 roughly 28 days following receipt of a single dose of a monovalent inactivated influenza A/H7N9 virus vaccine in individuals who previously received two intramuscular doses of a monovalent inactivated influenza A/H7N7 virus vaccine or are A/H7 vaccine-naïve.

The secondary objectives are 1. To assess study-vaccine related unsolicited non-serious adverse events following receipt of one dose of a monovalent inactivated influenza A/H7N9 virus vaccine in individuals who previously received two intramuscular doses of a monovalent inactivated influenza A/H7N7 virus vaccine or are A/H7 vaccine-naïve. 2. To assess new-onset chronic medical conditions following receipt of one dose of a monovalent inactivated influenza A/H7N9 virus vaccine in individuals who previously received two intramuscular doses of a monovalent inactivated influenza A/H7N7 virus vaccine or are A/H7 vaccine-naïve.3) To assess the serum HAI antibody responses against A/H7N9 at baseline and about 8 days following receipt of a single dose of a monovalent inactivated influenza A/H7N9 virus vaccine in individuals who previously received two intramuscular doses of a monovalent inactivated influenza A/H7N7 virus vaccine or are A/H7 vaccine-naïve. 4. To assess the serum neutralizing (Neut) antibody responses against A/H7N9 at baseline and roughly 8 and 28 days following receipt of a one dose of a monovalent inactivated influenza A/H7N7 virus vaccine or are A/H7 vaccine-naïve.

ELIGIBILITY:
Inclusion Criteria:

1. Provide written informed consent prior to initiation of any study procedures.
2. Are able to understand and comply with planned study procedures and be available for all study visits.
3. Are males or non-pregnant females, 19 to 50 years old, inclusive.
4. Are in good health*. *As determined by medical history and targeted physical examination, if indicated based on medical history, to evaluate acute or currently ongoing chronic medical diagnoses or conditions, defined as those that have been present for at least 90 days, that would affect the assessment of the safety of subjects or the immunogenicity of the study vaccination. Chronic medical diagnoses or conditions should be stable for the last 60 days. This includes no change in chronic prescription medication, dose, or frequency of as a result of deterioration of the chronic medical diagnosis or condition in the 60 days prior to enrollment. Any prescription change that is due to change of health care provider, insurance company, etc., or that is done for financial reasons, as long as in the same class of medication, will not be considered a deviation of this inclusion criterion. Any change in prescription medication due to improvement of a disease outcome, as determined by the site principal investigator or appropriate sub-investigator, will not be considered a deviation of this inclusion criterion. Subjects may be on chronic or as needed (prn) medications if, in the opinion of the site principal investigator or appropriate sub-investigator, they pose no additional risk to subject safety or assessment of reactogenicity and immunogenicity and do not indicate a worsening of medical diagnosis or condition. Similarly, medication changes subsequent to enrollment and the study vaccination are acceptable provided there was no deterioration in the subject's chronic medical condition that necessitated a medication change, and there is no additional risk to the subject or interference with the evaluation of responses to the study vaccination. Note: Topical, nasal, and inhaled medications (with the exception of inhaled corticosteroids as outlined in the Subject Exclusion Criteria (see Section 5.1.2), herbals, vitamins, and supplements are permitted.
5. Oral temperature is less than 100.0F.
6. Pulse is 50 to 115 bpm, inclusive.
7. Systolic blood pressure is 85 to 150 mmHg, inclusive.
8. Diastolic blood pressure is 55 to 95 mmHg, inclusive.
9. Women of childbearing potential** in sexual relationships with men must use an acceptable method of preventing conception*** from 30 days prior to 60 days after the study vaccination.

   **Not sterilized via tubal ligation, bilateral oophorectomy, hysterectomy or successful Essure® placement (permanent, non-surgical, non-hormonal sterilization) with documented radiological confirmation test at least 90 days after the procedure, and still menstruating or <1 year of the last menses if menopausal.

   ***Includes, but is not limited to, sexual abstinence, monogamous relationship with vasectomized partner who has been vasectomized for 180 days or more prior to the subject receiving the study vaccination, barrier methods such as condoms or diaphragms with spermicide or foam, effective intrauterine devices, NuvaRing®, and licensed hormonal methods such as implants, injectables or oral contraceptives ("the pill).
10. Women of childbearing potential must have a negative urine or serum pregnancy test within 24 hours prior to the study vaccination.
11. Received either two doses of an inactivated influenza A/H7N7 vaccine or one or two doses of placebo in DMID Protocol 07-0023 or have not received an influenza A/H7 vaccine.

Exclusion Criteria:

1. Have an acute illness*, as determined by the site principal investigator or appropriate sub-investigator, within 72 hours prior to the study vaccination.

   * An acute illness which is nearly resolved with only minor residual symptoms remaining is allowable if, in the opinion of the site principal investigator or appropriate sub-investigator, the residual symptoms will not interfere with the ability to assess safety parameters as required by the protocol.
2. Have any medical disease or condition that, in the opinion of the site principal investigator or appropriate sub-investigator, is a contraindication to study participation**.

   **Including acute or chronic medical disease or condition, defined as persisting for at least 90 days, that would place the subject at an unacceptable risk of injury, render the subject unable to meet the requirements of the protocol, or may interfere with the evaluation of responses or the subject's successful completion of this study.
3. Have immunosuppression as a result of an underlying illness or treatment, or use of anticancer chemotherapy or radiation therapy (cytotoxic) within 3 years prior to the study vaccination.
4. Have known active neoplastic disease or a history of any hematologic malignancy. Nonmelanoma skin cancers are permitted.
5. Have known human immunodeficiency virus (HIV), hepatitis B, or hepatitis C infection.
6. Have known hypersensitivity or allergy to eggs, egg or chicken protein, or other components of the study vaccine.
7. Have a history of severe reactions following previous immunization with licensed or unlicensed influenza virus vaccines.
8. Have a history of Guillain-Barré syndrome.
9. Have a history of alcohol or drug abuse within 5 years prior to the study vaccination.
10. Have any diagnosis, current or past, of schizophrenia, bipolar disease, or other psychiatric diagnosis that may interfere with subject compliance or safety evaluations.
11. Have been hospitalized for psychiatric illness, history of suicide attempt, or confinement for danger to self or others within 10 years prior to the study vaccination.
12. Have taken oral or parenteral (including intraarticular) corticosteroids of any dose within 30 days prior to the study vaccination.
13. Have taken high-dose*** inhaled corticosteroids within 30 days prior to the study vaccination****.

    ***High-dose defined as >840 mcg/day of beclomethasone dipropionate CFC or equivalent.

    ****Topical and nasal steroids are permissible.
14. Receipt or planned receipt of any licensed live vaccine, including seasonal influenza vaccine, within 30 days prior to 28 days after the study vaccination.
15. Receipt or planned receipt of any licensed inactivated vaccine, including seasonal influenza vaccine, within 14 days prior to 28 days after the study vaccination.
16. Received immunoglobulin or other blood products (with exception of Rho D immunoglobulin) within 90 days prior to the study vaccination.
17. Received an experimental agent***** within 30 days prior to the study vaccination, or expect to receive an experimental agent****** during the 6-month study-reporting period.

    *****Including vaccine, drug, biologic, device, blood product, or medication.

    ******Other than from participation in this study.
18. Are participating or plan to participate in another clinical study with an interventional agent during the 6-month study-reporting period.

    Note: Including licensed or unlicensed vaccine, drug, biologic, device, blood product, or medication.
19. Female subjects who are breastfeeding or plan to breastfeed at any given time from the study vaccination until 30 days after the study vaccination.
20. Blood donation or planned blood donation within 30 days prior to the study vaccination through 30 days after the last blood drawn for this study.

Ages: 19 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 27 (Actual)
Dates: Start 2016-01-12 (Actual); Primary Completion 2016-12-29 (Actual); Study Completion 2016-12-29 (Actual)

PRIMARY OUTCOMES:
Percent achieving HAI seroconversion against A/H7N9 antigen in A/H7N9 vaccine defined as either pre-vaccine HAI titer <1:10 and post-vaccine HAI titer > /= 1:40 or pre-vaccine HAI titer > /= 1:10 and minimum 4-fold rise in post-vaccine HAI antibody titer | Approximately 28 days after the A/H7N9 study vaccination.
Occurrence of solicited injection site and systemic reactogenicity events. | Time of the A/H7N9 study vaccination through 8 days after the A/H7N9 study vaccination.
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the A/H7N9 study vaccine. | Approximately 28 days after the A/H7N9 study vaccination.
Occurrence of study vaccine-related serious adverse events. | Time of the A/H7N9 study vaccination through approximately 6 months after the A/H7N9 study vaccination

SECONDARY OUTCOMES:
Percent achieve Neut seroconversion against A/H7N9 antigen in A/H7N9 vaccine, defined as either pre-vaccine Neut titer <1:10 and post-vaccine Neut titer > /= 1:40 or pre-vaccine Neut titer > /= 1:10 and min 4-fold rise in post-vaccine Neut antibody titer | Approximately 8 and 28 days after the A/H7N9 study vaccination.
Occurrence of study vaccine-related unsolicited non-serious adverse events. | Time of the A/H7N9 study vaccination through approximately 28 days after the A/H7N9 study vaccination.
Percentage of subjects achieving HAI seroconversion against the A/H7N9 antigen contained in the A/H7N9 study vaccine. | Approximately 8 days after A/H7N9 the study vaccination.
Percentage of subjects achieving a serum HAI antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the A/H7N9 study vaccine. | At baseline and approximately 8 days after the A/H7N9 study vaccination.
Percentage of subjects achieving a serum Neut antibody titer of 1:40 or greater against the A/H7N9 antigen contained in the A/H7N9 study vaccine. | At baseline and approximately 8 and 28 days after the A/H7N9 study vaccination.
Geometric Mean Titers of serum HAI and Neut antibodies against the A/H7N9 antigen contained in the A/H7N9 study vaccine. | At baseline and approximately 8 and 28 days after the A/H7N9 study vaccination.
Occurrence of new-onset chronic medical conditions. | Time of the A/H7N9 study vaccination through 6 months after the A/H7N9 study vaccination.

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine - Molecular Virology and Microbiology, Houston, Texas, United States

REFERENCES:
- [Derived] El Sahly HM, Atmar RL, Patel SM, Bellamy A, Liu L, Hong W, Zhu H, Guan Y, Keitel WA; DMID 13-0033 Vaccine Study Group. Safety and immunogenicity of an 8 year interval heterologous prime-boost influenza A/H7N7-H7N9 vaccination. Vaccine. 2019 May 1;37(19):2561-2568. doi: 10.1016/j.vaccine.2019.03.071. Epub 2019 Apr 4. PMID 30955980